CLINICAL TRIAL: NCT00199797
Title: Phase I Trial of huA33 Plus 5-fluorouracil (5-FU), Leucovorin and Oxaliplatin in Patients With Metastatic Colorectal Cancer
Brief Title: Phase I Trial of huA33 Plus Chemotherapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2003-005
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; huA33; antibody; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- huA33 antibody plus chemotherapy (Experimental): huA33 was administered intravenously over a period of 30 minutes once a week at a dose of 10 mg/m2 for 12 weeks.
  Starting on day 15 and continuing every second week, oxaliplatin, 5-fluorouracil (5-FU) and leucovorin were also administered.
  Oxaliplatin and leucovorin were given as infusions over 2 hours. Afterwards, patients received a bolus infusion of 5-FU intravenously followed by an infusion of 5-FU over 22 hours.
  The doses of oxaliplatin were 85mg/m2, leucovorin 200mg/m2, 400mg/m2 of 5-FU as a bolus infusion and 600mg/m2 as a continuous infusion.
  A complete treatment cycle consisted of 12 weeks. Patients were eligible to receive an additional cycle in the absence of dose-limiting toxicity (DLT), immunogenicity (huA33 human anti-human antibodies {HAHA}) and disease progression.
  Interventions: Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: huA33

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin was administered at 85 mg/m2 on day 2 of every 2 week regimen.
  Other Names: Eloxatin
Drug: 5-Fluorouracil — The dose of 5-FU was 400 mg/m2 IV bolus followed by continuous IV infusion at 600 mg/m2 over 22 hours on day 2 and day 3 of every 2 week regimen.
  Other Names: 5-FU
Drug: Leucovorin — Leucovorin was administered at a dose of 200mg/m2 on day 2 and day 3 of every 2 week regimen.
  Other Names: folinic acid
Drug: huA33 — huA33 was administered intravenously over a period of 30 minutes once a week at a dose of 10 mg/m2.

SUMMARY:
Although treatment for metastatic colorectal cancer has improved significantly over the recent years, it still remains a significant health problem representing the leading cancer by incidence in the United States of America. In the search for new therapies, monoclonal antibodies have been developed to specifically target human colon cancer cells. huA33 is an antibody that reacts with the A33 antigen which is produced by colorectal cancers. Prior studies have shown that administration of the huA33 antibody may delay the growth of tumor cells producing the specific antigen. Oxaliplatin and 5-fluorouracil (5-FU) are cytotoxic agents which are considered as standard treatment in metastatic colorectal cancer. Leucovorin (folinic acid) is a vitamin which enhances the effect of 5-FU. Eligible patients with advanced colorectal cancer will receive huA33 10 mg/m2 by intravenous (IV) infusion weekly for twelve weeks. Starting on Study Day 15 (week 3), 5-FU, leucovorin, and oxaliplatin will be administered every 2 weeks for 10 weeks. Patients will be evaluated weekly for toxicity. Blood samples will be obtained every week for hematology and serum biochemistry analysis and for determination of human anti-human antibodies (HAHA). In patients with measurable disease, tumors will be assessed by the appropriate scan at baseline and at the end of the thirteen week cycle. The primary objective of this study is to assess the safety of huA33 + 5-FU + leucovorin + oxaliplatin. The secondary objective is to measure the immunogenicity of huA33 when given in combination with 5-FU plus leucovorin and oxaliplatin and to document tumor responses.

DETAILED DESCRIPTION:
Purpose of the Research Study:

huA33 is an antibody that reacts with the A33 antigen which is produced by colorectal cancers. Prior studies have shown that application of the huA33 antibody may delay the growth of tumor cells producing the respective antigen.

Oxaliplatin and 5-FU are cytotoxic agents which are considered as standard treatment in metastatic colorectal cancer. Leucovorin is a vitamin which enhances the effect of 5-FU.

The primary purpose of this study is to determine whether the combination huA33 plus oxaliplatin, 5-FU and leucovorin is safe and what side effects occur.

Description of Research Procedures:

The first step is to determine whether or not patients are eligible for participation in the study. Apart from general blood tests and x-ray studies needed, this involves testing with regard to some special requirements:

* Three tests of stool to determine if it is positive for blood.
* Women of childbearing age must have a negative pregnancy test.
* If patients ever had a treatment with similar substances like huA33 before, a blood sample needs to be tested for antibodies that may have developed against huA33.

After eligibility is established, huA33 will be administered intravenously over a period of 30 minutes once a week at a dose of 10 mg/m2. Starting on day 15 and continuing every second week, oxaliplatin, 5-FU and leucovorin are administered. Oxaliplatin and leucovorin will be given as infusions over 2 hours. Afterwards patients will receive a bolus infusion of 5-FU intravenously followed by an infusion of 5-FU over 22 hours.

The doses of oxaliplatin will be 85mg/m2, leucovorin 200mg/m2, 400mg/m2 of 5-FU as a bolus infusion and 600mg/m2 as a continuous infusion. A complete treatment cycle consists of 12 weekly treatment days.

Patients will have an interview with their doctor and a physical examination before the first day of treatment and before each therapy. Standard blood tests as well as special blood tests to measure a possible reaction of the immune system to the huA33 antibody will be done weekly and before the treatment is started. The amount of blood to be drawn will be 20-30 ml during one cycle of the study.

X-rays and/or CT scans to measure the extent of the disease will be done at the start and at week 13, which is considered to be the first day of the next cycle. Patients may continue with this treatment for up to 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for enrollment if they fulfill all of the following criteria:

1. Metastatic colorectal cancer.
2. Histologically or cytologically proven colorectal cancer.
3. Expected survival of at least 4 months.
4. Not more than 2 different pretreatment regimens.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
6. Within the 2 weeks prior to the first dose of huA33, the following vital laboratory parameters:

   Lab Parameter Range
   * Neutrophil count ≥ 1.5 x 10E9/L
   * Platelet count ≥ 150 x 10E9/L
   * Serum bilirubin ≤ 2 mg/dL
   * Creatinine clearance >50 ml/ min
7. Age ≥ 18 years.
8. Able and willing to give valid written informed consent.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

1. Untreated active metastatic disease to the central nervous system defined as new or enlarging lesions on CT or MRI.
2. Surgery or radiotherapy of brain metastases within 3 months prior to the first dose of huA33.
3. Metastatic disease involving > 50% of liver volume.
4. Other serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders.
5. Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing (6 weeks for nitrosoureas).
6. Previous treatment with oxaliplatin.
7. Previous treatment with huA33 monoclonal antibody or antibody fragment.

   a. Positive huA33 HAHA titer - defined as greater than 3 standard deviations above the mean patient normal range by Biacore analysis.
8. Concomitant treatment with systemic corticosteroids. Topical or inhalational corticosteroids are permitted.
9. Known HIV, Hepatitis B or C positivity.
10. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
11. Lack of availability of the patient for clinical and laboratory follow-up assessment.
12. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing.
13. Pregnancy or breastfeeding.
14. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-04-18 (Actual); Primary Completion 2006-11-08 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Renner, MD, Principal Investigator — Universitätsspital Zürich, Switzerland; Alexander Knuth, MD, Principal Investigator — Universitätsspital Zürich, Switzerland; Elke Jäger, MD, Principal Investigator — Krankenhaus Nordwest, Germany
Locations (2):
- Krankenhaus Nordwest, Frankfurt, Germany
- UniversitaetsSpital Zuerich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | huA33 Antibody Plus Chemotherapy
Started | 20
Completed | 17
Not Completed | 3
Not completed — Progressive Disease | 1
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of huA33.
Groups:
- huA33 Antibody Plus Chemotherapy: huA33 was administered intravenously over a period of 30 minutes once a week at a dose of 10 mg/m2 for 12 weeks.
  Starting on day 15 and continuing every second week, oxaliplatin, 5-fluorouracil (5-FU) and leucovorin were also administered.
  Oxaliplatin and leucovorin were given as infusions over 2 hours. Afterwards, patients received a bolus infusion of 5-FU intravenously followed by an infusion of 5-FU over 22 hours.
  The doses of oxaliplatin were 85mg/m2, leucovorin 200mg/m2, 400mg/m2 of 5-FU as an bolus infusion and 600mg/m2 as a continuous infusion.
  A complete treatment cycle consisted of 12 weeks. Patients were eligible to receive an additional cycle in the absence of dose-limiting toxicity (DLT), immunogenicity (huA33 human anti-human antibodies {HAHA}) and disease progression.
Arm/Group | huA33 Antibody Plus Chemotherapy
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 66 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 2
  Germany | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by the Number of Patients With Treatment Emergent Adverse Events (TEAEs), Grade 3 TEAEs, TEAEs Resulting in Death, TEAEs Related to Treatment and Serious TEAEs in Patients With Metastatic Colorectal Cancer.
Description: Patients were evaluated weekly for toxicity. Blood samples were obtained every week for hematology and serum biochemistry analysis. All adverse events, which occurred after the signing of informed consent were documented in the case report form. Toxicity was evaluated according to the National Cancer Institute CTCAE Scale (Version 3.0). All AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 13.1 and classified by MedDRA system organ class (SOC) and preferred term. Treatment emergent adverse events (TEAEs) are any adverse events occurring or worsening after the first administration of study drug.
Time Frame: up to 26 weeks
Population: All patients who received at least one dose of huA33.
Measure: Count of Participants; unit: Participants
Arm/Group | huA33 Antibody Plus Chemotherapy
Number analyzed (Participants) | 20
Participants
  Number of patients with treatment emergent adverse events | 20
  Number of patients with treatment emergent adverse events Grade 3 or above | 17
  Number of patients with treatment emergent adverse events which resulted in death | 1
  Number of patients with treatment emergent adverse events related to treatment | 18
  Number of patients with serious adverse events | 11

2. Secondary Outcome: Immunogenicity of huA33 as Measured by the Number of Patients With Human Anti-human Antibodies (HAHA) When Given huA33 Together With Oxaliplatin and 5-FU Plus Leucovorin in Patients With Metastatic Colorectal Cancer.
Description: Serum samples were taken at baseline and prior to each administration of huA33.The samples were analyzed by surface plasmon resonance technology using a BIACORE 2000 instrument. All sera were analyzed at the end of the study. Patient serum was considered HAHA positive if the response unit (RU) value at a serum dilution of 1:100 exceeded a cutoff value, defined as the mean inter-patient baseline RU value + 3x the standard deviation (SD) of negative control sera at a serum dilution of 1:100. Results were reported as either positive or negative.
Time Frame: up to 26 weeks
Population: All patients who received at least one dose of huA33.
Measure: Count of Participants; unit: Participants
Groups:
- huA33 Antibody Plus Chemotherapy: huA33 was administered intravenously over a period of 30 minutes once a week at a dose of 10 mg/m2 for 12 weeks.
  Starting on day 15 and continuing every second week, oxaliplatin,5-fluorouracil (5-FU) and leucovorin were also administered.
  Oxaliplatin and leucovorin were given as infusions over 2 hours. Afterwards, patients received a bolus infusion of 5-FU intravenously followed by an infusion of 5-FU over 22 hours.
  The doses of oxaliplatin were 85mg/m2, leucovorin 200mg/m2, 400mg/m2 of 5-FU as an bolus infusion and 600mg/m2 as a continuous infusion.
  A complete treatment cycle consisted of 12 weeks. Patients were eligible to receive an additional cycle in the absence of dose-limiting toxicity (DLT), immunogenicity (huA33 human anti-human antibodies {HAHA}) and disease progression.
Arm/Group | huA33 Antibody Plus Chemotherapy
Number analyzed (Participants) | 20
Participants
  Patients with positive HAHA response | 6
  Patients with negative HAHA response | 14

3. Secondary Outcome: Tumor Response in Patients With Metastatic Colorectal Cancer Receiving huA33, Oxaliplatin and 5-FU Plus Leucovorin.
Description: Tumor response was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) (Therasse P et al. J Natl Cancer Inst 92: 205-216 2000) at baseline and at the end of each cycle.
  Per RECIST, target lesions were categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria.
Time Frame: up to 26 weeks
Population: Patients who received huA33 and were evaluable for response. One patient was not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | huA33 Antibody Plus Chemotherapy
Number analyzed (Participants) | 19
Participants
  Complete Response | 1
  Partial Response | 7
  Stable Disease | 4
  Progressive Disease | 7

ADVERSE EVENTS:
Time Frame: up to 26 weeks
Description: All adverse events which occurred after signing informed consent were documented in the source records and on the respective case report form, regardless of the assumption of a causal relationship. Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Scale (Version 3.0).Treatment emergent adverse events (TEAEs) are any adverse events occurring or worsening after the first administration of study drug.
Groups:
- huA33 Antibody Plus Chemotherapy: huA33 was administered intravenously over a period of 30 minutes once a week at a dose of 10 mg/m2 for 12 weeks.
  Starting on day 15 and continuing every second week, oxaliplatin,5-fluorouracil (5-FU) and leucovorin were also administered.
  Oxaliplatin and leucovorin were given as infusions over 2 hours. Afterwards patients received a bolus infusion of 5-FU intravenously followed by an infusion of 5-FU over 22 hours.
  The doses of oxaliplatin were 85mg/m2, leucovorin 200mg/m2, 400mg/m2 of 5-FU as a bolus infusion and 600mg/m2 as a continuous infusion.
  A complete treatment cycle consisted of 12 weeks. Patients were eligible to receive an additional cycle in the absence of dose-limiting toxicity (DLT), immunogenicity (huA33 human anti-human antibodies {HAHA}) and disease progression.
Arm/Group | huA33 Antibody Plus Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | huA33 Antibody Plus Chemotherapy (N=20)
Sudden death (General disorders) | 1
Chills (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Pyrexia (General disorders) | 2
Hypersensitivity (Immune system disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Performance status decreased (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Arterial thrombosis limb (Vascular disorders) | 1
Catheter placement (Surgical and medical procedures) | 1
Chemotherapy (Surgical and medical procedures) | 1
Device related infection (Infections and infestations) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | huA33 Antibody Plus Chemotherapy (N=20)
Neutropenia (Blood and lymphatic system disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Bradycardia (Cardiac disorders) | 4
Dyspnoea exertional (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 3
Nausea (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 4
Dysgeusia (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 9
Mucosal inflammation (General disorders) | 6
Pyrexia (General disorders) | 4
Pain (General disorders) | 4
Chills (General disorders) | 2
Asthenia (General disorders) | 2
Oedema peripheral (General disorders) | 2
Drug hypersensitivity (Immune system disorders) | 3
Nasopharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Weight decreased (Investigations) | 4
Blood creatinine increased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Respiratory rate increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Polyneuropathy (Nervous system disorders) | 9
Headache (Nervous system disorders) | 5
Sleep disorder (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 5
Pruritis (Skin and subcutaneous tissue disorders) | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 7
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No